CLINICAL TRIAL: NCT03973255
Title: Efficacy Of Biofeedback Training And Whole Body Vibration Therapy In Vestibular Rehabilitation Of Unilateral Vestibular Weakness
Brief Title: Whole Body Vibration In Vestibular Rehabilitation
Acronym: WBV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, Fazıl Necdet Ardıç, Prof.Dr.Fazıl Necdet Ardıç, Pamukkale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1
Record Dates: First submitted 2019-06-01; First posted 2019-06-04 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Vestibular Disease
Keywords: Vestibular rehabilitation; Vestibular weakness; Whole Body Vibration; Biofeedback; Posturography
MeSH Terms: conditions — Vestibular Diseases | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Home based vestibular rehabilitation program (Placebo Comparator): Home-based vestibular rehabilitation program including vestibular adaptation exercises, oculomotor exercises, static and dynamic balance exercises was given to each group in the form of a booklet. All exercises were demonstrated and performed first time at hospital under supervision. Booklet with descriptions and pictures of each exercise were given to patients in order to enable them to perform exercises at home. Vestibular rehabilitation exercises were prescribed as once daily with 10 repetitions at home for one month and wanted to mark a chart if the exercises were performed daily. A diary was used to monitor adherence with the program.
  Interventions: Behavioral: Rehabilitation
- Biofeedback training (Active Comparator): Biofeedback training was performed five days a week during a month for 20 minutes for a total of 20 sessions with Tetrax ® (Sunlight Medical Ltd) static posture analysis device. Biofeedback training including "catch, speedball, sky ball, gotcha" exercises which requires following a visual target during weight transfer movements, capturing fast-moving objects by changing the center of gravity or quickly escaping from incoming objects, were applied to the patients in biofeedback training. There is a 30 seconds pause between each exercise.
  Interventions: Behavioral: Rehabilitation
- Whole body vibration (Active Comparator): Whole body vibration training was also performed five days a week during a month for 20 minutes for a total of 20 sessions with Power Plate Pro 5 (MDD CE 0086). In whole body vibration, single leg, squat and deep squat positions were applied respectively with 35 Hz frequency, including rest periods of 30 seconds between each application.
  Interventions: Behavioral: Rehabilitation

INTERVENTIONS:
Behavioral: Rehabilitation — Posturography, Whole body vibration

SUMMARY:
The aim of this study was to compare the efficacy of home based vestibular rehabilitation program, posturographic biofeedback training and whole body vibration therapy on balance, fall risk, functional mobility, vertigo symptom severity and functions in patients with unilateral vestibular weakness.

DETAILED DESCRIPTION:
A total of 90 patients who were diagnosed as unilateral vestibular weakness were included in this prospective randomized controlled study. They were randomized into three groups each consisting of 30 patients. Home based vestibular rehabilitation program was given to all groups. Fall risk yielded by posturography, Berg balance scale, Timed Up-and-Go test, vertigo visual analogue scale and Dizziness Handicap Inventory were used for comparison.

ELIGIBILITY:
Inclusion Criteria:

Adult patients who had unilateral vestibular weakness and persistent dizziness at least two months after acute period were included Bithermal caloric test showing hyporesponsiveness higher than 30% or unresponsiveness of the horizontal canal of the affected ear accepted as unilateral vestibular weakness.

Exclusion Criteria:

Bilateral vestibular weakness, Recurrent vestibulopathy, Benign paroxysmal positional vertigo, Concomitant neurological or psychiatric disease, Severe visual or auditory impairments and orthopedic problems in the lower extremities

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-03-13 (Actual); Primary Completion 2019-01-31 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
fall risk | 30 days
  fall risk yielded by static posturography
Berg balance scale | 30 days
  BBS consists of 14 tasks that are each scored on a scale of 0-4, for a total possible score of 56, indicating no identified balance difficulties. Scoring is on a 5-point ordinal scale with 0 indicating an inability to complete the task and 4 as independent in completing the task.
Timed Up-and-Go | 30 days
  TUG is a balance and gait index which requires subjects to rise from an armchair, walk 3 m at a normal and safe pace, turn around, walk back to the chair and sit-down. The time required to complete this task is measured in seconds.
vertigo visual analogue scale | 30 days
  A vertically oriented 10 cm line was used for VAS, where "no vertigo" corresponds to the bottom of the line and "the worst vertigo that they could imagine" corresponds to the top of the line. Patients were instructed to place a mark on the 10-cm vertical line according to severity of their vertigo.
Dizziness Handicap Inventory | 30 days
  The DHI has 25 items, sub-grouped into three domains: functional, emotional, and physical. There are three closed-form answers where patients may check one of the following: yes, sometimes and no with the corresponding scored as 4/2/0. It is possible to use both the total score and the scores of the three subscales separately.

CONTACTS AND LOCATIONS:
Overall Officials: Fazıl N Ardıç, MD, Principal Investigator — Pamukkale University
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No